CLINICAL TRIAL: NCT00520377
Title: Pilot Study on Safety and Efficacy of MD05 in Comparison With Beta-TCP in Patients Undergoing Sinus Floor Augmentation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Scil Technology GmbH (Industry)
Collaborators: FGK Clinical Research GmbH (Industry)
Responsible Party: Björn Capsius, Scil Technology GmbH
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Scil-MD05-C01; Sinus Lift Study
Record Dates: First submitted 2007-08-23; First posted 2007-08-24 (Estimated); Last update posted 2008-04-23 (Estimated); Status verified 2008-04

CONDITIONS: Alveolar Ridge Augmentation
Keywords: Sinus Lift Surgery; Sinus Floor Augmentation; Insufficient Bone Height

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): MD05
  Interventions: Drug: MD05
- 2 (Active Comparator): Beta-TCP and autologous bone
  Interventions: Device: Beta-TCP and autologous bone

INTERVENTIONS:
Drug: MD05 — recombinant human GDF-5 coated onto beta-tricalcium phosphate
  Arms: 1
Device: Beta-TCP and autologous bone — beta-tricalcium phosphate and autologous bone
  Arms: 2

SUMMARY:
The primary objective is the area of newly formed bone (%) as assessed by histomorphometry with either MD05 or beta-TCP.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring two-stage unilateral maxillary sinus floor augmentation (sinus lift) in case of insufficient bone height in the area of the posterior maxilla, prior to insertion of dental implants
* Residual bone height at the site of planned implantation > 1 mm and < 5 mm
* Male and female outpatients, 18 to 75 years old
* Female patients must be infertile (either sterilized or postmenopausal). If a patient's menopausal status at screening is uncertain, levels of follicle stimulating hormone (FSH) should be determined. Patients with an FSH level > 25 IU/l and absence of menstrual bleeding > 6 months will satisfy the definition of postmenopausal status.
* Patient has given informed consent.

Exclusion Criteria:

* Women of childbearing potential, lactating women
* Participation in another clinical study within 30 days prior to study start
* Previous participation in this study
* Last dental extraction (maxilla, posterior to canine) within the last 3 months
* Failed sinus lift surgery and previous eradictive maxillary sinus surgery
* Simultaneously bilateral sinus lift
* Legal incompetence or restricted legal competence
* Alcoholism, drug dependency, smoking
* Acute or chronic infection at the application site, e.g., sinusitis
* Known infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV)
* Severe allergic rhinitis which requires permanent medication (Rosenlicht 1999)
* Known intolerance of or hypersensitivity to beta-TCP or rhGDF﷓-5
* Presence of local or systemic malignant disease or history of local or systemic malignant disease in the past 5 years
* Patients requiring chemo- or radiotherapy
* Previous or current radiotherapy of the head
* Chronic liver disorder
* Impaired renal function
* Uncontrolled, insulin-dependent diabetes mellitus
* Clinically relevant symptoms of thyroid dysfunction
* Severe hypertension (RRdiast > 110 mmHg);
* Clinically relevant cardiovascular disease
* Systemic bone disease or illness having influence on bone metabolism,
* Clinically relevant blood coagulation disorder,
* Leukopenia < 3.500 leukocytes/µL
* Previous or current treatment with systemic corticosteroids
* Previous or current therapy with drugs having any influence on bone metabolism
* Previous or current treatment with immunosuppressant medication

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2005-01; Primary Completion 2007-12 (Actual); Study Completion 2008-05 (Estimated)

PRIMARY OUTCOMES:
Area of newly formed mineralised bone tissue (%) as assessed by histomorphometry. | Within 4 months after surgery

SECONDARY OUTCOMES:
evidence of uncompromised healing | January 2008

CONTACTS AND LOCATIONS:
Overall Officials: Wilfried Wagner, Prof Dr Dr, Principal Investigator — Universitätsklinikum Mainz
Locations (9):
- Germany (9):
  - Universitätsklinik Erlangen, Erlangen, Bavaria
  - Praxis Dr. Gath, München, Bavaria
  - IPI München GmbH, München, Bavaria
  - Praxis Dr. Schmidinger, Seefeld, Bavaria
  - Universitätsklinik Düsseldorf, Düsseldorf, North Rhine-Westphalia
  - Klinikum der Universität Mainz, Mainz, Rheinland Pflaz
  - Universitätsklinikum Schleswig Holstein, Kiel, Schleswig-Holstein
  - Charité Universitätsmedizin Berlin, Berlin, State of Berlin
  - Helios Klinik, Erfurt, Thuringia